CLINICAL TRIAL: NCT00003518
Title: Phase II Study of Paclitaxel Plus Gemcitabine in Refractory Germ Cell Tumors
Brief Title: Paclitaxel Plus Gemcitabine in Treating Patients With Refractory Metastatic Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000066562; E9897
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel plus gemcitabine in treating patients with refractory metastatic germ cell tumors that have not responded to surgery or chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the effect of gemcitabine plus paclitaxel on response rate, duration of remission, and survival in patients with refractory germ cell tumors. II. Evaluate the toxic effects of this regimen in these patients.

OUTLINE: Patients receive paclitaxel IV over 1 hour followed by gemcitabine IV over 30 minutes on days 1, 8, and 15 of each 4 week course. Treatment is repeated for a maximum of six courses in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for 2 years, every 6 months for 3 years, then annually thereafter.

PROJECTED ACCRUAL: Approximately 44 patients will be accrued over 19 months for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or serologically confirmed metastatic germ cell neoplasm (gonadal or extragonadal primary) that cannot be cured with either surgery or chemotherapy Seminomas, nonseminomas, or ovarian germ cell tumors allowed If histologically confirmed, requires one or more of the following: Metastatic lesions on chest x-ray or CT scan Rising serum HCG or AFP If only evidence of progressive disease, then two additional consecutive determinations must exhibit serologic progression Only eligible if alternative causes for increased serum levels are absent Failed initial cisplatin combination chemotherapy (generally bleomycin/etoposide/cisplatin, cisplatin/etoposide, cisplatin/vinblastine, or similar regimens) Failed and demonstrated progressive disease following the administration of at least one "salvage" regimen for advanced germ cell neoplasms Failed no more than three prior regimens defined as: 25% increase in the product of perpendicular diameters of measurable tumor masses during prior therapy, new lesions OR Increasing AFP or HCG Disease progression during initial induction chemotherapy or with primary mediastinal nonseminomatous germ cell tumors can be treated with paclitaxel plus gemcitabine as second-line therapy (initial salvage chemotherapy)

PATIENT CHARACTERISTICS: Age: 15 and over Performance status: ECOG 0-2 Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT no greater than 4 times normal Bilirubin no greater than 2 mg/dL Renal: Creatinine no greater than 2.5 mg/dL Other: No active uncontrolled infection Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: At least 3 weeks since major surgery and recovered Other: At least 1 week since prior intravenous antibiotics No concurrent intravenous antibiotics

Ages: 15 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 1999-01-25 (Actual); Primary Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence H. Einhorn, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (19):
- United States (18):
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Einhorn LH, Brames MJ, Juliar B, Williams SD. Phase II study of paclitaxel plus gemcitabine salvage chemotherapy for germ cell tumors after progression following high-dose chemotherapy with tandem transplant. J Clin Oncol. 2007 Feb 10;25(5):513-6. doi: 10.1200/JCO.2006.07.7271. PMID 17290059
- [Result] Hinton S, Catalano P, Einhorn LH, Loehrer PJ Sr, Kuzel T, Vaughn D, Wilding G. Phase II study of paclitaxel plus gemcitabine in refractory germ cell tumors (E9897): a trial of the Eastern Cooperative Oncology Group. J Clin Oncol. 2002 Apr 1;20(7):1859-63. doi: 10.1200/JCO.2002.07.158. PMID 11919245